CLINICAL TRIAL: NCT04229797
Title: The Efficacy of Mandibular First Molar Distalization Using Extra Radicular Miniscrews in Class III Patients: A Randomized Clinical Trial
Brief Title: Mandibular First Molar Distalization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Khaled Makhlouf, Associate researcher NRC, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MakhloufOrth
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Class III Malocclusion
Keywords: Class III malocclusion; Mandibular buccal shelf; Mini-screws; Extra-radicular mini-screws; Distalization; Temporary Anchorage device
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparator (Active Comparator): Extraction of the unerupted third molars before distalization of mandibular first molar using Mandibular buccal shelf mini-screws.
  Interventions: Procedure: Mandibular distalization using extra-radicular miniscrews
- Intervention (Experimental): Leaving the unerupted third molars and distalizing using Mandibular buccal shelf mini-screws.
  Interventions: Procedure: Mandibular distalization using extra-radicular miniscrews

INTERVENTIONS:
Procedure: Mandibular distalization using extra-radicular miniscrews — Distalization of the Mandibular first molars using mandibular buccal shelf mini-screws in the presence of unerupted third molars

SUMMARY:
A clinical study to test the capability of the mini-screws inserted in the Mandibular buccal shelf area as an anchorage unit to distalize mandibular first molar for correction of mild to moderate Class III cases. The second aim was to detect if there is a difference in the amount of distalization in the presence of unerupted mandibular third molars, using the same technique.

DETAILED DESCRIPTION:
Class III malocclusion in adults is one of the most complex malocclusions in clinical orthodontics. For adults, the ideal treatment option for Class III malocclusion is accomplished either by camouflage treatment in mild to moderate cases or orthognathic surgery in severe cases. Camouflage treatment for Class III malocclusion comprises three main techniques; Class III elastics, mandibular first molar distalization, or extraction of mandibular first premolars. Mandibular first molar distalization via the use of skeletal anchorage has the problem of increased failure rate of the inter-radicular temporary anchorage devices (TADs). Accordingly, a randomized clinical trial using extra radicular TADs in the Mandibular buccal shelf area was designed in the current research aiming to test the efficacy of such a technique in inducing mandibular molar distalization with decreased failure rate, and whether the presence of unerupted mandibular third molars will affect the distalization movement or not.

ELIGIBILITY:
Inclusion Criteria:

* Class III dental incisal relation.
* Dental canine and molar relation not more than half unit Class III.
* Presence of unerupted mandibular third molars on both sides.
* Skeletal Class I or mild Class III.
* Full Permanent dentition.
* Medically free subjects.

Exclusion Criteria:

* Patients with systemic diseases or neuromuscular disorders.
* Retroclined lower incisors.
* Sever skeletal dysplasia.
* Patients with periodontal disease.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dental effect | 6 months
  Amount of first mandibular molar distalization (mm) in the two groups, A cephalometric of pre and post distalization digital cephalograms will be traced, landmarks and reference lines will be determined; skeleto-dental and soft tissue measurements will be performed using Quick-Ceph program .
  Digital models of pre and post distalization will be superimposed and measured for dental changes using Anatomage program.

SECONDARY OUTCOMES:
Skeletal and soft tissue effect | 6 months
  Skeletal and soft tissue changes post distalization, A cephalometric of pre and post distalization digital cephalograms will be traced, landmarks and reference lines will be determined; skeleto-dental and soft tissue measurements will be performed using Quick-Ceph program.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No